CLINICAL TRIAL: NCT04947150
Title: Optimizing an mHealth Intervention to Change Food Purchasing Behaviors for Cancer Prevention
Acronym: EatWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Meghan Butryn, Associate Professor of Psychology, Drexel University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R21CA252933 (NIH); 1R21CA252933 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-01 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a 2x2x2x2 design. There are four factors, each with two levels: ON vs OFF.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LOCATION TRIGGERED MESSAGING (Experimental): Weekly message is triggered when arriving at grocery store.
  Interventions: Behavioral: Location-triggered notification
- COACH MONITORING (Experimental): Coaches view grocery purchases via web portal, send weekly messages about purchases they observe, and conduct three brief phone calls to discuss purchases.
  Interventions: Behavioral: Coach monitoring
- BENEFITS OF CHANGE (Experimental): Attend an extra workshop session and three phone calls to identify and reflect on benefits of dietary change. Content added to standard weekly messages about benefits of change.
  Interventions: Behavioral: Reflections on benefits of change
- HOUSEHOLD SUPPORT (Experimental): An adult household member attends one workshop session and three phone calls with the index participant. This household member receives weekly text messages for 20 weeks about program goals and ways to support the index participant.
  Interventions: Behavioral: Household support

INTERVENTIONS:
Behavioral: Location-triggered notification — If participants are randomized to have this component ON, the app will send the notification when the participant's smartphone is within a 50-meter "geofence" around designated grocery stores. No more than one notification will be sent per week. Mindfulness of program goals in the moment of decision making is expected to facilitate program-consistent food purchasing behaviors. Participants assigned to have location-triggered message delivery OFF will receive their weekly "recommendations and reminders" messages at standard times throughout the week. The content of the messages will not differ according to whether this component is ON vs. OFF.
  Arms: LOCATION TRIGGERED MESSAGING
Behavioral: Reflections on benefits of change — Participants will reflect on anticipated benefits of purchasing healthy foods, consistent with motivational interviewing and self-determination theory. Message content will be personalized as follows: During the initial workshop, all participants will complete an exercise identifying benefits of healthy eating that are important to them. Message content will then be programmed to be personalized according to anticipated rewards important to that participant. Participants assigned to have this intervention component OFF will not have content about anticipated benefits of change added to any messages.
  Arms: BENEFITS OF CHANGE
Behavioral: Coach monitoring — Coaches will monitor participant food purchases via a dashboard for viewing purchase data, and send messages designed to provide feedback and enhance supportive accountability for program goals. The messages will provide reinforcement for purchases consistent with program goals and express concern for areas in which adherence is low. Participants assigned to have this component OFF will not receive these extra messages or phone calls, and their food purchases will only be viewed by research staff for research outcome assessment purposes.
  Arms: COACH MONITORING
Behavioral: Household support — If participants are assigned to have household support ON, one adult in the household will receive weekly text messages designed to elicit support for changing food purchases. In addition, the index participant and household member will be invited to participate in one extra workshop session and three brief coaching calls focused on household support. If participants are assigned to have this OFF, household members will have no program involvement.
  Arms: HOUSEHOLD SUPPORT

SUMMARY:
Dietary intake is a powerful, modifiable factor that influences cancer risk. Unfortunately, most adults in the U.S. find it difficult to adhere to dietary guidelines for cancer prevention. One promising pathway for improving dietary adherence is to target grocery shopping habits, i.e., foods purchased for consumption at home. Two-thirds of daily food intake is sourced from or eaten in the home, so improving the quality of the home food environment should improve overall diet quality. When healthy foods are purchased and unhealthy foods are not, minimal self-control is needed to make healthy eating choices in the home. At the point of purchase, it is difficult to resist the temptation of palatable foods, but interventions might facilitate healthy choices by promoting dietary goal salience in real-time while grocery shopping, enhancing motivation to make and sustain changes to the diet, and increasing household support and accountability for healthy food purchasing. The proposed study will enroll adults who have low adherence to cancer prevention dietary recommendations. All participants will attend a nutrition education workshop conducted via Zoom. For 20 weeks, all participants also will receive once weekly reminders and recommendations for food purchasing via an app. The study will experimentally test four additional intervention components: location-triggered messages, coaching monitoring of food purchases, benefit of change content, and household member involvement. The preliminary aim of the study is to assess feasibility and acceptability of the intervention components. The primary aim of the study is to quantify the effect of each intervention component, individually and in combination, on dietary intake (assessed with 24-hour food recalls). The overarching goal of this project is to optimize this mHealth intervention, which can be tested in the future in a fully powered clinical trial.

ELIGIBILITY:
Inclusion criteria

* 18 years or older
* Fluent in English
* Low adherence to cancer prevention dietary guidelines, operationalized as a score of ≤ 2 out of 4 using the National Cancer Institute method for assessing adherence to World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) lifestyle recommendations. This three-level scoring system (meeting/partially meeting/not meeting each recommendation) includes 4 items specific to diet. Participants must score equal or less than 2, meaning that they are fully meeting recommendations for no more than 2 of the 4 dietary recommendations.
* Performs the majority of the household's food shopping, and do so at stores that can passively stream item-level data from a store loyalty card to the Information Machine API (e.g., Walmart, Target, ShopRite, Wegman's, etc.)
* Has a smartphone with iOS or Android operating system that is compatible with the program app
* Lives in a household with at least one other adult who consents to being randomized to possibly receive messages on his/her own cell phone through the program app

Exclusion criteria

* Medical condition or psychiatric condition (e.g., active substance abuse, eating disorder) that may limit appropriateness of or ability to comply with program dietary recommendations
* Planning to enroll in another lifestyle modification program in the next 6 months
* Bariatric surgery history
* Currently pregnant or breastfeeding or planning to become pregnant in the next 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan L Butryn, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Butryn ML, Hagerman CJ, Crane NT, Ehmann MM, Forman EM, Milliron BJ, Simone NL. A Proof-of-Concept Pilot Test of a Behavioral Intervention to Improve Adherence to Dietary Recommendations for Cancer Prevention. Cancer Control. 2023 Jan-Dec;30:10732748231214122. doi: 10.1177/10732748231214122. PMID 37950612
- [Derived] Horgan OZ, Crane NT, Forman EM, Milliron BJ, Simone NL, Zhang F, Butryn ML. Optimizing an mHealth Intervention to Change Food Purchasing Behaviors for Cancer Prevention: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 24;11(6):e39669. doi: 10.2196/39669. PMID 35749216

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The four experimental intervention components are each provided to 50% of participants.
Groups:
- Condition 1: Location triggered messaging - OFF, Benefits of change - OFF, Coach monitoring - OFF, Household support - OFF.
- Condition 2: Location triggered messaging - ON, Benefits of change - OFF, Coach monitoring - OFF, Household support - OFF.
- Condition 3: Location triggered messaging - ON, Benefits of change - ON, Coach monitoring - OFF, Household support - OFF.
- Condition 4: Location triggered messaging - ON, Benefits of change - ON, Coach monitoring - ON, Household support - OFF.
- Condition 5: Location triggered messaging - ON, Benefits of change - ON, Coach monitoring - ON, Household support - ON.
- Condition 6: Location triggered messaging - ON, Benefits of change - ON, Coach monitoring - OFF, Household support - ON.
- Condition 7: Location triggered messaging - ON, Benefits of change - OFF, Coach monitoring - ON, Household support - ON.
- Condition 8: Location triggered messaging - ON, Benefits of change - OFF, Coach monitoring - OFF, Household support - ON.
- Condition 9: Location triggered messaging - ON, Benefits of change - OFF, Coach monitoring - ON, Household support - OFF.
- Condition 10: Location triggered messaging - OFF, Benefits of change - ON, Coach monitoring - OFF, Household support - OFF.
- Condition 11: Location triggered messaging - OFF, Benefits of change - ON, Coach monitoring - ON, Household support - OFF.
- Condition 12: Location triggered messaging - OFF, Benefits of change - ON, Coach monitoring - ON, Household support - ON.
- Condition 13: Location triggered messaging - OFF, Benefits of change - ON, Coach monitoring - OFF, Household support - ON.
- Condition 14: Location triggered messaging - OFF, Benefits of change - OFF, Coach monitoring - ON Household support - OFF.
- Condition 15: Location triggered messaging - OFF, Benefits of change - OFF, Coach monitoring - OFF, Household support - ON.
- Condition 16: Location triggered messaging - OFF, Benefits of change - OFF, Coach monitoring - ON, Household support - ON.
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
Started | 4 | 7 | 2 | 2 | 7 | 2 | 5 | 2 | 3 | 5 | 6 | 2 | 5 | 2 | 4 | 4
Wave 1 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1 | 2 | 1 | 2 | 2
Wave 2 | 2 | 5 | 1 | 0 | 5 | 0 | 3 | 1 | 1 | 3 | 4 | 1 | 3 | 1 | 2 | 2
Completed | 4 | 7 | 1 | 2 | 7 | 0 | 4 | 2 | 3 | 5 | 5 | 1 | 5 | 1 | 4 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Total
Number analyzed (Participants) | 4 | 7 | 2 | 2 | 7 | 2 | 5 | 2 | 3 | 5 | 6 | 2 | 5 | 2 | 4 | 4 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (19.5) | 53.6 (11.0) | 47.5 (27.6) | 53.0 (11.3) | 46.7 (14.9) | 36.0 (15.6) | 52.4 (15.3) | 45.0 (9.9) | 35.0 (7.0) | 44.8 (9.9) | 48.3 (11.4) | 39.5 (17.7) | 56.0 (8.4) | 40.5 (17.7) | 43.3 (20.0) | 42.3 (12.1) | 47.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 2 | 2 | 7 | 1 | 4 | 2 | 3 | 5 | 6 | 1 | 5 | 2 | 4 | 4 | 57
  Male | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 6
  Not Hispanic or Latino | 4 | 7 | 1 | 2 | 7 | 2 | 5 | 2 | 2 | 5 | 5 | 2 | 5 | 1 | 3 | 3 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 1 | 3 | 4 | 0 | 2 | 0 | 2 | 0 | 21
  White | 2 | 5 | 1 | 1 | 3 | 1 | 4 | 0 | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 2 | 33
  More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Education level [Count of Participants; unit: Participants]
  Completed postgraduate or professional degree | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 2 | 0 | 3 | 1 | 18
  Graduated from college | 2 | 2 | 1 | 0 | 4 | 2 | 2 | 1 | 1 | 2 | 3 | 1 | 2 | 2 | 1 | 3 | 29
  Completed some college | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 12
  Completed senior high | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Household size [Count of Participants; unit: Participants]
  Two | 1 | 3 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 3 | 1 | 3 | 1 | 3 | 1 | 24
  Three | 0 | 3 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 15
  Four | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 16
  Five or more | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 7
Grocery shopping frequency [Count of Participants; unit: Participants]
  Less than once per week | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 6
  Once per week | 3 | 2 | 2 | 0 | 4 | 0 | 4 | 1 | 0 | 4 | 2 | 1 | 3 | 1 | 1 | 1 | 29
  Twice per week | 0 | 3 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 4 | 0 | 1 | 0 | 2 | 1 | 18
  More than twice per week | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 9
Weight [Mean (Standard Deviation); unit: pounds] | 242.8 (31.2) | 199.3 (32.8) | 145.0 (35.4) | 168.5 (6.4) | 205.7 (50.7) | 190.0 (11.3) | 173.4 (44.7) | 208.5 (128.0) | 177.3 (35.0) | 180.8 (43.7) | 211.3 (53.9) | 216.0 (76.4) | 168.4 (36.8) | 152.0 (53.7) | 166.0 (58.2) | 164.3 (37.0) | 188.7 (47.8)
Body Mass Index [Mean (Standard Deviation); unit: kg^m2] | 40.0 (5.1) | 33.9 (7.4) | 24.3 (3.3) | 31.3 (1.9) | 36.2 (8.5) | 29.8 (1.8) | 28.1 (7.8) | 38.0 (18.9) | 30.7 (5.6) | 31.2 (6.0) | 36.1 (9.1) | 34.8 (16.3) | 28.0 (5.2) | 24.7 (7.2) | 28.0 (9.6) | 29.5 (5.7) | 32.1 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: 1a. Dietary Intake: ASA24 (Fiber)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in grams of fiber per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: Participants were randomly assigned to whether each of the four conditions were "on" (location triggered messaging, coach monitoring, benefits of change, and household report). Change across time for each outcome are reported for each condition and for the full sample.
  The Ns reported here are smaller than the full trial sample because only Wave 1 participants completed the ASA-24. Results here only include Wave 1 participants.
Measure: Mean (Standard Error); unit: grams/day
Groups:
- Coach Monitoring - ON: Coaches view grocery purchases via web portal, send weekly messages about purchases they observe, and conduct three brief phone calls to discuss purchases.
  Coach monitoring: Coaches will monitor participant food purchases via a dashboard for viewing purchase data, and send messages designed to provide feedback and enhance supportive accountability for program goals. The messages will provide reinforcement for purchases consistent with program goals and express concern for areas in which adherence is low. Participants assigned to have this component OFF will not receive these extra messages or phone calls, and their food purchases will only be viewed by research staff for research outcome assessment purposes.
- Coach Monitoring - OFF: Participants did not receive coach monitoring
- Benefits of Change - ON: Attend an extra workshop session and three phone calls to identify and reflect on benefits of dietary change. Content added to standard weekly messages about benefits of change.
  Reflections on benefits of change: Participants will reflect on anticipated benefits of purchasing healthy foods, consistent with motivational interviewing and self-determination theory. Message content will be personalized as follows: During the initial workshop, all participants will complete an exercise identifying benefits of healthy eating that are important to them. Message content will then be programmed to be personalized according to anticipated rewards important to that participant. Participants assigned to have this intervention component OFF will not have content about anticipated benefits of change added to any messages.
- Benefits of Change - OFF: Participants did not receive a benefits of change intervention.
- Location Triggered Messaging - ON: Weekly message is triggered when arriving at grocery store.
  Location-triggered notification: If participants are randomized to have this component ON, the app will send the notification when the participant's smartphone is within a 50-meter "geofence" around designated grocery stores. No more than one notification will be sent per week. Mindfulness of program goals in the moment of decision making is expected to facilitate program-consistent food purchasing behaviors. Participants assigned to have location-triggered message delivery OFF will receive their weekly "recommendations and reminders" messages at standard times throughout the week. The content of the messages will not differ according to whether this component is ON vs. OFF.
- Location Triggered Messaging - OFF: Participants did not receive location triggered messaging intervention
- Household Support - ON: An adult household member attends one workshop session and three phone calls with the index participant. This household member receives weekly text messages for 20 weeks about program goals and ways to support the index participant.
  Household support: If participants are assigned to have household support ON, one adult in the household will receive weekly text messages designed to elicit support for changing food purchases. In addition, the index participant and household member will be invited to participate in one extra workshop session and three brief coaching calls focused on household support. If participants are assigned to have this OFF, household members will have no program involvement.
- Household Support - OFF: Participants did not receive the household support intervention.
- Full Sample: The total sample, includes all conditions
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
grams/day
  0 weeks (baseline) | 18.45 (2.12) | 18.17 (2.39) | 15.89 (2.31) | 20.73 (2.10) | 16.30 (2.45) | 20.32 (2.05) | 18.90 (2.25) | 17.72 (2.08) | 18.31 (1.53)
  20 weeks (post-treatment) | 18.51 (2.91) | 14.19 (3.28) | 16.98 (3.2) | 15.72 (2.89) | 14.50 (3.37) | 18.20 (2.82) | 18.40 (3.09) | 14.30 (2.86) | 16.35 (2.11)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .255, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA were used

2. Primary Outcome: 1b. Primary Outcome: Dietary Intake ASA24 (Fruit/Veg)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in number of cups of fruits and vegetables per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Cups/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
Cups/day
  0 weeks (baseline) | 1.86 (.40) | 2.63 (.44) | 2.40 (.43) | 2.09 (.39) | 2.33 (.46) | 2.16 (.38) | 2.41 (.42) | 2.08 (.39) | 2.25 (.29)
  20 weeks (post-treatment) | 2.70 (.58) | 2.15 (.65) | 2.67 (.63) | 2.18 (.57) | 2.10 (.66) | 2.75 (.56) | 2.69 (.61) | 2.16 (.56) | 2.42 (.42)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .560, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

3. Primary Outcome: 1c. Primary Outcome: Dietary Intake ASA24 (Red Meat)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in ounces of red meat consumed per week.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: oz/week
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
oz/week
  0 weeks (baseline) | 10.10 (4.40) | 8.98 (4.95) | 4.10 (4.79) | 14.98 (4.35) | 4.35 (5.08) | 14.72 (4.25) | 13.13 (4.66) | 5.95 (4.31) | 9.54 (3.18)
  10 weeks (post-treatment) | 3.71 (2.06) | 8.39 (2.32) | 8.23 (2.24) | 3.87 (2.04) | 4.36 (2.38) | 7.74 (1.99) | 3.91 (2.18) | 8.19 (2.02) | 6.05 (1.49)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .319, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

4. Primary Outcome: 1d. Primary Outcome: Dietary Intake ASA24 (Processed Meat)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in ounces of processed meat consumed per week.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: oz/week
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
oz/week
  0 weeks (baseline) | 325.95 (109.76) | 216.18 (123.43) | 282.69 (119.44) | 259.44 (108.47) | 278.05 (126.79) | 264.09 (106.06) | 371.70 (116.32) | 170.44 (107.53) | 271.07 (79.20)
  10 weeks (post-treatment) | 97.34 (31.24) | 49.79 (35.13) | 74.12 (33.99) | 73.01 (30.87) | 87.96 (37.08) | 59.17 (30.18) | 72.10 (33.10) | 75.03 (30.60) | 73.56 (22.54)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .032, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

5. Primary Outcome: 1e. Primary Outcome: Dietary Intake ASA24 (Added Sugars)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in grams of added sugars consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
grams/day
  0 weeks (baseline) | 41.82 (8.72) | 31.16 (9.81) | 28.30 (9.49) | 44.67 (8.62) | 34.25 (10.08) | 38.72 (8.43) | 40.93 (9.24) | 32.04 (8.55) | 36.49 (6.30)
  20 weeks (post-treatment) | 25.63 (7.20) | 17.11 (8.10) | 11.84 (7.84) | 30.91 (7.12) | 21.93 (8.32) | 20.81 (6.96) | 21.94 (7.63) | 20.81 (7.05) | 21.37 (5.20)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .044, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

6. Primary Outcome: 1f. Primary Outcome: Dietary Intake ASA24 (Sodium)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in mg of sodium consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
mg/day
  0 weeks (baseline) | 730.13 (86.00) | 571.33 (81.16) | 647.89 (83.99) | 653.57 (79.51) | 663.92 (82.30) | 637.53 (82.16) | 676.85 (81.75) | 624.61 (83.57) | 650.73 (59.94)
  20 weeks (post-treatment) | 440.77 (99.20) | 323.50 (93.62) | 323.24 (96.88) | 441.03 (91.71) | 343.04 (94.94) | 421.24 (94.77) | 353.12 (94.30) | 411.15 (96.40) | 382.14 (65.68)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .010, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated Measures ANOVA

7. Primary Outcome: 1g. Primary Outcome: Dietary Intake ASA24 (Fat)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in grams of saturated fat consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
grams/day
  0 weeks (baseline) | 9.27 (1.15) | 7.91 (1.08) | 9.05 (1.12) | 8.13 (1.06) | 9.86 (1.10) | 7.32 (1.10) | 9.47 (1.09) | 7.71 (1.12) | 8.59 (.76)
  20 weeks (post-treatment) | 4.92 (1.06) | 3.59 (1.00) | 3.76 (1.04) | 4.74 (.98) | 4.17 (1.02) | 4.34 (1.02) | 3.67 (1.01) | 4.84 (1.03) | 4.25 (.70)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .073, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

8. Primary Outcome: 1h. Primary Outcome: Dietary Intake ASA24 (Sugar-Sweetened Beverages)
Description: In Wave 1, the primary outcome will be change from 0-20 weeks in dietary intake of the major food categories from the American Institute for Cancer Research guidelines. Self-reported dietary recalls will be completed for three days at baseline and week 20 using the Automated Self Administered 24-hour food recall (ASA-24). This table reports the change in oz of sugar sweetened beverages consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: oz/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 14 | 28
oz/day
  0 weeks (baseline) | 17.29 (6.85) | 17.39 (6.46) | 21.44 (6.69) | 13.24 (6.33) | 24.64 (6.55) | 10.04 (6.54) | 19.79 (6.51) | 14.90 (6.66) | 17.34 (4.53)
  20 weeks (post-treatment) | 18.72 (5.09) | 6.84 (4.81) | 14.38 (4.97) | 11.18 (4.71) | 7.71 (4.87) | 17.85 (4.86) | 10.55 (4.84) | 15.01 (4.95) | 12.78 (3.37)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .872, ANOVA — The reported p-value reflects the change across time for the full (Wave 1) sample; Repeated measures ANOVA

9. Primary Outcome: 2a: Dietary Intake: DHQ-III (Fiber)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in grams of fiber per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: Participants were randomly assigned to whether each of the four conditions were "on" (location triggered messaging, coach monitoring, benefits of change, and household report). Change across time for each outcome are reported for each condition and for the full sample.
  The Ns reported here are smaller than the full trial sample because only Wave 2 participants completed the DHQ-III. Results here only include Wave 2 participants.
Measure: Mean (Standard Error); unit: grams/day
Groups:
- Coach Monitoring - OFF: Participants did not receive the coach monitoring intervention.
- Benefits of Change - OFF: Participants did not receive the benefits of change intervention.
- Location-Triggered Messaging - OFF: Participants did not receive the location triggered messaging intervention.
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
grams/day
  0 weeks (baseline) | 16.94 (2.41) | 16.83 (2.28) | 18.38 (2.36) | 15.38 (2.23) | 18.98 (2.31) | 14.78 (2.31) | 15.56 (2.29) | 18.21 (2.34) | 16.88 (1.60)
  20 weeks (post-treatment) | 20.18 (3.90) | 18.24 (3.68) | 20.65 (3.81) | 17.78 (3.60) | 21.37 (3.73) | 17.05 (3.73) | 18.79 (3.71) | 19.63 (3.79) | 19.21 (2.58)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .145, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated Measures ANOVA

10. Primary Outcome: 2b. Dietary Intake: DHQ-III (Fruits/Veg)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in cups of fruits and vegetables per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: cups/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
cups/day
  0 weeks (baseline) | 2.56 (.42) | 2.93 (.39) | 3.06 (.41) | 4.23 (.39) | 3.31 (.40) | 2.17 (.40) | 2.61 (.40) | 2.88 (.41) | 2.74 (.28)
  20 weeks (post-treatment) | 3.09 (.69) | 3.35 (.66) | 3.47 (.68) | 2.97 (.64) | 3.84 (.66) | 2.60 (.66) | 3.26 (.66) | 3.18 (.67) | 3.22 (.46)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .173, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

11. Primary Outcome: 2c. Dietary Intake: DHQ-III (Red Meat)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in oz of red meat consumed per week.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: oz/week
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
oz/week
  0 weeks (baseline) | 4.43 (.82) | 3.49 (.77) | 3.01 (.80) | 4.90 (.76) | 3.88 (.78) | 4.04 (.78) | 3.13 (.78) | 4.79 (.80) | 3.96 (.54)
  20 weeks (post-treatment) | 2.66 (.70) | 3.03 (.66) | 2.48 (.69) | 3.21 (.65) | 2.77 (.67) | 2.92 (.67) | 2.46 (.67) | 3.23 (.68) | 2.84 (.47)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .012, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

12. Primary Outcome: 2d. Dietary Intake: DHQ-III (Processed Meat)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in oz of processed meat consumed per week.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: oz/week
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
oz/week
  0 weeks (baseline) | 165.20 (57.26) | 133.88 (54.04) | 103.41 (55.92) | 195.66 (52.94) | 59.94 (54.80) | 239.14 (54.70) | 133.67 (54.43) | 165.40 (55.64) | 149.54 (37.91)
  20 weeks (post-treatment) | 40.72 (12.12) | 48.04 (11.43) | 35.75 (11.83) | 53.01 (11.20) | 31.86 (11.60) | 56.89 (11.58) | 25.92 (11.52) | 62.84 (11.77) | 44.38 (8.02)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .008, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

13. Primary Outcome: 2e. Dietary Intake: DHQ-III (Added Sugars)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in grams of added sugars consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
grams/day
  0 weeks (baseline) | 28.37 (5.01) | 24.53 (4.73) | 28.35 (4.89) | 24.55 (4.63) | 30.27 (4.79) | 22.62 (4.78) | 26.53 (4.76) | 23.37 (4.87) | 26.45 (3.32)
  20 weeks (post-treatment) | 16.98 (4.84) | 14.06 (4.57) | 16.69 (4.73) | 14.35 (4.48) | 15.01 (4.64) | 16.04 (4.63) | 13.38 (4.60) | 17.67 (4.71) | 15.52 (3.21)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

14. Primary Outcome: 2f. Dietary Intake: DHQ-III (Sodium)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in mg of sodium consumed per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
mg/day
  0 weeks (baseline) | 730.13 (86.00) | 571.33 (81.16) | 647.89 (83.99) | 653.57 (79.51) | 663.92 (82.30) | 637.53 (82.16) | 676.85 (81.75) | 624.61 (83.57) | 650.73 (59.94)
  20 weeks (post-treatment) | 440.77 (99.20) | 323.50 (93.62) | 323.24 (96.88) | 441.03 (91.71) | 343.04 (94.94) | 421.24 (94.77) | 353.12 (94.30) | 411.15 (96.40) | 382.14 (65.68)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

15. Primary Outcome: 2g. Dietary Intake: DHQ-III (Fat)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in grams of saturated fat per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
grams/day
  0 weeks (baseline) | 9.27 (1.15) | 7.91 (1.08) | 9.05 (1.12) | 8.13 (1.06) | 9.86 (1.10) | 7.32 (1.10) | 9.47 (1.09) | 7.71 (1.12) | 8.59 (.76)
  20 weeks (post-treatment) | 4.92 (1.06) | 3.59 (1.00) | 3.76 (1.04) | 4.74 (.98) | 4.17 (1.02) | 4.34 (1.02) | 3.67 (1.01) | 4.84 (1.03) | 4.25 (.70)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

16. Primary Outcome: 2h. Dietary Intake: DHQ-III (Sugar-Sweetened Beverages)
Description: In Wave 2, the Diet History Questionnaire (DHQ-III) will be used instead of food recalls to assess dietary intake. This table reports the change in ounces of sugar-sweetened beverages per day.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 9
Measure: Mean (Standard Error); unit: grams/day
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 16 | 18 | 17 | 17 | 34
grams/day
  0 weeks (baseline) | 17.29 (6.85) | 17.39 (6.46) | 21.44 (6.69) | 13.24 (6.33) | 24.64 (6.55) | 10.04 (6.54) | 19.79 (6.51) | 14.90 (6.66) | 17.34 (4.53)
  20 weeks (post-treatment) | 18.72 (5.09) | 6.84 (4.81) | 14.38 (4.97) | 11.18 (4.71) | 7.71 (4.87) | 17.85 (4.86) | 10.55 (4.84) | 15.01 (4.95) | 12.78 (3.37)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .382, ANOVA — The reported p-value reflects the change across time for the full (Wave 2) sample; Repeated measures ANOVA

17. Secondary Outcome: Goal Salience
Description: Goal salience while grocery shopping was measured using an investigator-developed self-report questionnaire. Participants rated 3 questions pertaining to salience of health goals during grocery shopping on a sliding scale from 0 (not at all) to 100 (very much): Scores on these three items were averaged to compute a global Goal Salience total score (range = 0-100), with higher scores indicating higher goal salience.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: Participants were randomly assigned to whether each of the four conditions were "on" (location triggered messaging, coach monitoring, benefits of change, and household report). Change across time for each outcome are reported for each condition and for the full sample.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Location Triggered Messaging - OFF: Participants did not receive the location triggered messaging intervention.
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 56.62 (4.62) | 53.35 (4.32) | 57.97 (4.46) | 53.99 (4.16) | 53.80 (4.42) | 58.16 (4.31) | 59.02 (4.21) | 53.94 (4.47) | 55.98 (3.02)
  10 weeks (mid-treatment) | 71.96 (4.22) | 72.04 (3.94) | 74.40 (4.06) | 69.60 (3.79) | 74.52 (4.03) | 69.48 (3.93) | 71.93 (3.84) | 72.07 (4.07) | 72.00 (2.75)
  20 weeks (post-treatment) | 66.58 (3.96) | 69.23 (3.70) | 70.67 (3.82) | 65.14 (3.56) | 70.88 (3.79) | 64.93 (3.70) | 69.61 (3.61) | 66.20 (3.83) | 67.90 (2.58)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated Measures ANOVA

18. Secondary Outcome: Supportive Accountability
Description: Supportive accountability was measured using 5 items adapted from the Perceptions of Accountability Scale (Chhabria et al., 2020). Participants rated 5 items (e.g., "I feel accountable to others for meeting my dietary goals") on a sliding scale from 0 (not at all) to 100 (very much). Scores on the 5 items were averaged to produce a global Supportive Accountability total score (range 0-100), with higher scores indicating higher perceived supportive accountability to others for dietary/healthy eating goals.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 54.89 (5.11) | 44.23 (4.77) | 51.69 (4.93) | 47.42 (4.60) | 48.39 (4.89) | 50.73 (4.77) | 46.62 (4.66) | 52.40 (4.94) | 49.56 (3.33)
  10 weeks (mid-treatment) | 52.82 (4.99) | 50.53 (4.66) | 57.13 (4.81) | 46.22 (4.49) | 50.86 (4.78) | 52.49 (4.66) | 49.55 (4.55) | 53.80 (4.82) | 51.67 (3.26)
  20 weeks (post-treatment) | 49.42 (4.84) | 43.19 (4.52) | 49.20 (4.67) | 43.41 (4.36) | 49.20 (4.63) | 43.41 (4.52) | 42.50 (4.41) | 50.11 (4.68) | 46.31 (3.16)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .178, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

19. Secondary Outcome: Autonomous Motivation
Description: Motivation for healthy eating was measured using 10 items adapted from the Treatment Self-Regulation Questionnaire (Levesque et al., 2007). Using the question stem "The reason I would follow a healthy diet is...", participants rated items on a scale from 1 (not at all true) to 7 (very true). Six items were averaged to create a subscale of autonomous Motivation for healthy eating (range 1-7), with higher scores on each subscale indicated higher Autonomous Motivation.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 6.32 (.15) | 6.48 (.14) | 6.34 (.14) | 6.46 (.13) | 6.43 (.14) | 6.37 (.14) | 6.42 (.13) | 6.38 (.14) | 6.40 (.10)
  10 weeks (Midtreatment) | 6.32 (.22) | 6.03 (.20) | 5.96 (.21) | 6.39 (.20) | 6.22 (.21) | 6.13 (.20) | 6.11 (.20) | 6.24 (.21) | 6.18 (.14)
  20 weeks (Post-Treatment) | 6.09 (.15) | 6.28 (.14) | 6.09 (.14) | 6.27 (.13) | 6.32 (.14) | 6.05 (.14) | 6.44 (.13) | 5.93 (.14) | 6.18 (.10)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .081, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

20. Secondary Outcome: External Motivation
Description: Motivation for healthy eating was measured using 10 items adapted from the Treatment Self-Regulation Questionnaire (Levesque et al., 2007). Using the question stem "The reason I would follow a healthy diet is...", participants rated items on a scale from 1 (not at all true) to 7 (very true). Four items were averaged to create the subscale of external Motivation for healthy eating (range 1-7). Higher scores on each subscale indicated higher external motivation for healthy eating.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (Baseline) | 2.82 (.28) | 2.75 (.26) | 2.89 (.27) | 2.68 (.25) | 2.82 (.27) | 2.75 (.26) | 2.71 (.25) | 2.86 (.27) | 2.78 (.18)
  10 weeks (Midtreatment) | 3.19 (.29) | 2.74 (.27) | 2.88 (.28) | 3.05 (.26) | 2.88 (.28) | 3.05 (.27) | 2.72 (.27) | 3.21 (.28) | 2.96 (.19)
  20 weeks (Post-Treatment) | 2.95 (.28) | 2.44 (.26) | 2.74 (.27) | 2.65 (.25) | 2.80 (.27) | 2.58 (.26) | 2.32 (.25) | 3.06 (.27) | 2.69 (.18)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .343, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

21. Secondary Outcome: Social Support (Encouragement)
Description: Participants responded to 10 items adapted from the Sallis Social Support for Diet Questionnaire (Sallis et al., 1987). Using the question stem "The other adult(s) in my household...", participants rated items on a scale from 1 (none) to 5 (very often), with 6 indicating "Not Applicable" (N/A; recoded as 1). Five items were summed to measure encouragement of healthy eating (e.g., "complimented me on changing my eating habits"; range 5-25), with higher scores indicating higher encouragement. This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (Baseline) | 14.05 (.90) | 12.51 (.84) | 13.64 (.87) | 12.91 (.81) | 13.31 (.86) | 13.24 (.84) | 12.39 (.82) | 14.16 (.87) | 13.28 (.59)
  10 weeks (Midtreatment) | 14.16 (1.03) | 14.46 (.96) | 14.66 (.99) | 13.95 (.92) | 14.54 (.98) | 14.08 (.96) | 14.46 (.94) | 14.16 (.99) | 14.31 (.67)
  20 weeks (Post-Treatment) | 13.65 (1.14) | 14.14 (1.07) | 14.02 (1.10) | 13.78 (1.03) | 13.24 (1.09) | 14.55 (1.07) | 14.66 (1.04) | 13.14 (1.11) | 13.90 (12.40)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .369, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

22. Secondary Outcome: Social Support (Discouragement)
Description: Participants completed the Sallis Social Support for Diet Questionnaire (Sallis et al., 1987). Using the question stem "The other adult(s) in my household...", participants rated items on a scale from 1 (none) to 5 (very often). 6 indicated "Not Applicable," which was recoded as 1 (none). Five items (e.g., "ate unhealthy foods in front of me") were summed to create the Discouragement of Healthy Eating subscale (range 5-25); higher scores indicated higher discouragement.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (Baseline) | 13.64 (.99) | 13.37 (.92) | 13.55 (.95) | 13.46 (.89) | 13.42 (.95) | 13.59 (.92) | 13.64 (.90) | 13.37 (.95) | 13.51 (.64)
  10 weeks (Midtreatment) | 12.64 (.90) | 11.56 (.84) | 11.43 (.87) | 12.76 (.81) | 11.03 (.86) | 13.16 (.84) | 11.28 (.82) | 12.91 (.87) | 12.10 (.59)
  20 weeks (Post-Treatment) | 12.71 (1.01) | 12.10 (.94) | 11.91 (.97) | 12.90 (.91) | 11.26 (.97) | 13.55 (.94) | 11.88 (.92) | 12.93 (.98) | 12.40 (.66)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .055, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

23. Secondary Outcome: Quality of Household Relationship
Description: Quality of the household relationship was measured using 5 items adapted from the Relationship Assessment Scale (Hendrick, 1988). Items assessed the quality of their relationship with the person who served as their household support partner in the Eatwell program (e.g., "How well does this person meet your needs") on a scale from 1 (Low) to 5 (High). Scores on the 5 items were averaged to calculate a Relationship Quality total score (range 1-5); higher scores indicated higher perceived relationship quality.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline
Population: Participants were randomly assigned to whether each of the four conditions were "on" (location triggered messaging, coach monitoring, benefits of change, and household report). Baseline scores are reported for each condition and for the full sample.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale | 4.10 (.13) | 4.41 (.13) | 4.30 (.13) | 4.21 (.13) | 4.19 (.13) | 4.32 (.13) | 4.33 (.13) | 4.18 (.13) | 4.25 (.72)

24. Secondary Outcome: Weight History
Description: Weight history was measured using an investigator developed questionnaire. Participants answered the following question about weight history in the past 6 months: "Which of these statements best describe what has happened to your weight during the past 6 months?" Answer choices included: (1) My weight has stayed the same; (2) I've been losing weight; (3) I've been gaining weight; or (4) My weigh has fluctuated a lot.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 weeks (Baseline)
Population: as for outcome 23
Measure: Number; unit: count of participants
Groups:
- Coach Monitoring Condition - ON: Coaches view grocery purchases via web portal, send weekly messages about purchases they observe, and conduct three brief phone calls to discuss purchases.
  Coach monitoring: Coaches will monitor participant food purchases via a dashboard for viewing purchase data, and send messages designed to provide feedback and enhance supportive accountability for program goals. The messages will provide reinforcement for purchases consistent with program goals and express concern for areas in which adherence is low. Participants assigned to have this component OFF will not receive these extra messages or phone calls, and their food purchases will only be viewed by research staff for research outcome assessment purposes.
- Coaching Monitoring Condition - OFF: Participants did not receive the coach monitoring intervention
Arm/Group | Coach Monitoring Condition - ON | Coaching Monitoring Condition - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
count of participants
  My weight has stayed about the same | 11 | 14 | 16 | 9 | 12 | 13 | 13 | 12 | 25
  I've been losing weight | 2 | 5 | 4 | 3 | 3 | 4 | 5 | 2 | 7
  I've been gaining weight | 14 | 6 | 6 | 14 | 10 | 10 | 10 | 10 | 20
  My weight has fluctuated a lot | 4 | 6 | 5 | 5 | 5 | 5 | 3 | 7 | 10

25. Secondary Outcome: Dietary Restraint
Description: Dietary restraint was measured using the Three Factor Eating Questionnaire (Cappelleri et al., 2009). For items #1-20, participants rated statements on a 4-point Likert scale from 1 (definitely true) to 4 (definitely false; reverse coded). Item 21 assessed overall restraint on an 8-point scale from 1 (no restraint) to 8 (total restraint), recoded such that 1-2=1; 3-4=2; 5-6=3; and 7-8=4 (so that all items ranged 1-4). Six items were summed to calculate a Restraint score (range = 6-24); higher scores indicated more restraint.
  This pilot study used a factorial design, with 16 conditions and ~4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (Baseline) | 15.98 (.60) | 14.71 (.55) | 15.21 (.57) | 15.49 (.55) | 15.12 (.58) | 15.57 (.55) | 14.77 (.55) | 15.92 (.57) | 15.34 (.39)
  10 weeks (Midtreatment) | 16.82 (.62) | 16.45 (.57) | 17.04 (.59) | 16.22 (.56) | 17.00 (.60) | 16.27 (.57) | 16.65 (.57) | 16.61 (.59) | 16.63 (.40)
  20 weeks (Post-Treatment) | 16.57 (.65) | 17.05 (.60) | 16.80 (.62) | 16.82 (.59) | 17.37 (.62) | 16.24 (.60) | 17.12 (.59) | 16.50 (.62) | 16.81 (.42)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

26. Secondary Outcome: Uncontrolled Eating
Description: Uncontrolled eating was measured using the subscale of the Three Factor Eating Questionnaire - 21 item (Cappelleri et al., 2009). Responses ranged from 1 (definitely true) to 4 (definitely false). Items were reverse coded and summed to calculate an uncontrolled eating (range = 6-24), with higher scores indicating higher uncontrolled eating.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 20.03 (1.28) | 19.45 (1.20) | 19.47 (1.23) | 20.02 (1.25) | 19.37 (1.23) | 20.11 (1.19) | 20.63 (1.17) | 18.86 (1.24) | 19.74 (.84)
  10 weeks (mid-treatment) | 18.80 (1.11) | 18.13 (1.04) | 18.83 (1.07) | 18.10 (1.00) | 18.07 (1.06) | 18.86 (1.04) | 18.90 (1.01) | 18.03 (1.07) | 18.46 (.73)
  20 weeks (post-treatment) | 18.49 (1.17) | 17.91 (1.09) | 17.49 (1.12) | 18.90 (1.05) | 18.43 (1.11) | 17.97 (1.09) | 18.48 (1.06) | 17.91 (1.13) | 18.20 (.76)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .079, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

27. Secondary Outcome: Emotional Eating
Description: Emotional eating was measured using the subscale of the Three Factor Eating Questionnaire - 21 item (Cappelleri et al., 2009). Responses ranged from 1 (definitely true) to 4 (definitely false). Six were reverse coded and summed to calculate an emotional eating (range = 6-24), with higher scores indicating higher emotional eating.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0 (Baseline), 10 (Midtreatment), 20 weeks (Posttreatment)
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 14.43 (1.23) | 12.94 (1.15) | 13.21 (1.19) | 14.14 (1.11) | 12.98 (1.18) | 14.36 (1.15) | 13.08 (1.12) | 14.26 (1.19) | 13.67 (.80)
  10 weeks (mid-treatment) | 14.26 (1.07) | 12.87 (1.00) | 13.29 (1.03) | 13.83 (.96) | 13.46 (1.02) | 13.66 (1.00) | 13.19 (.97) | 13.93 (1.03) | 13.56 (.70)
  20 weeks (post-treatment) | 13.47 (1.14) | 13.04 (1.07) | 12.69 (1.10) | 13.82 (1.03) | 13.43 (1.09) | 13.08 (1.07) | 12.61 (1.04) | 13.90 (1.11) | 13.25 (.75)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .581, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

28. Secondary Outcome: Dietary Intake - FFQ (Guideline 1)
Description: A 13-item Food Frequency Questionnaire was adapted from similar measures (Rifas-Shiman et al., 2001). To measure intake for guideline 1 (i.e., fruits, vegetables, whole grains, and bean/ legumes ), participants rated how frequently they consumed these categories (4 items) during an average week over the past month (0=Never, 1=less than once per week, 2=once per week, 3=2-4 times/week, 4=nearly daily/daily, 5=greater than twice per day). A total guideline 1 score was calculated as the average of responses to the 4 items (range 0-5), where higher scores indicate more frequently eating fruits, vegetables, whole grains, and beans/legumes. This study used a factorial design, with 16 conditions (with ~4 participants) and was designed to collapse across conditions (i.e., comparing 8 conditions where factor is ON to 8 OFF conditions). Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0, 10, 20 weeks
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 2.71 (.16) | 2.58 (.15) | 2.74 (.16) | 2.56 (.15) | 2.79 (.15) | 2.51 (.15) | 2.60 (.15) | 2.70 (.16) | 2.65 (.11)
  20 weeks (post-treatment) | 3.48 (.20) | 3.08 (.18) | 3.39 (.19) | 3.17 (.18) | 3.36 (.19) | 3.19 (.18) | 3.25 (.18) | 3.31 (.19) | 3.28 (.13)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

29. Secondary Outcome: Dietary Intake - FFQ (Guideline 2)
Description: A 13-item Food Frequency Questionnaire was adapted from similar measures (Rifas-Shiman et al., 2001). To measure intake for guideline 2 (i.e., processed foods high in fat, starches, sugars), participants rated how frequently they consumed foods from these categories (6 items) during an average week over the past month (0=Never, 1=less than once per week, 2=once per week, 3=2-4 times/week, 4=nearly daily/daily, 5=greater than twice per day). A total guideline 2 score was calculated as the average of responses to the 6 items (range 0-5), where higher scores indicate more frequently eating processed foods. This study used a factorial design, with 16 conditions (with ~4 participants) and was designed to collapse across conditions (i.e., comparing 8 conditions where factor is ON to 8 OFF conditions). Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0, 10, 20 weeks
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 2.41 (.17) | 2.10 (.16) | 2.20 (.16) | 2.30 (.15) | 2.23 (.16) | 2.28 (.16) | 2.27 (.15) | 2.24 (.16) | 2.25 (.11)
  20 weeks (post-treatment) | 1.43 (.16) | 1.33 (.15) | 1.22 (.15) | 1.54 (.14) | 1.23 (.15) | 1.53 (.15) | 1.29 (.15) | 1.47 (.15) | 1.38 (.10)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

30. Secondary Outcome: Dietary Intake - FFQ (Guideline 3)
Description: A 13-item Food Frequency Questionnaire was adapted from similar measures (Rifas-Shiman et al., 2001). To measure intake for guideline 3 (i.e., red and processed meat), participants rated how frequently they consumed these categories (2 items) during an average week over the past month (0=Never, 1=less than once per week, 2=once per week, 3=2-4 times/week, 4=nearly daily/daily, 5=greater than twice per day). A total guideline 3 score was calculated as the average of responses to the 2 items (range 0-5), where higher scores indicate more frequently eating red and processed meats. This study used a factorial design, with 16 conditions (with ~4 participants) and was designed to collapse across conditions (i.e., comparing 8 conditions where factor is ON to 8 OFF conditions). Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0, 10, 20 weeks
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 1.82 (.19) | 1.98 (.17) | 1.68 (.18) | 2.12 (.17) | 1.77 (.18) | 2.02 (.17) | 1.84 (.17) | 1.98 (.18) | 1.90 (.12)
  20 weeks (post-treatment) | 1.11 (.16) | 1.08 (.15) | .91 (.16) | 1.28 (.15) | .95 (.15) | 1.24 (.15) | .93 (.15) | 1.26 (.16) | 1.09 (.11)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

31. Secondary Outcome: Dietary Intake - FFQ (Guideline 4)
Description: A 13-item Food Frequency Questionnaire was adapted from similar measures (Rifas-Shiman et al., 2001). To measure intake for guideline 4 (i.e., sugar-sweetened drinks), participants rated how frequently they consumed these drinks (1 item) during an average week over the past month (0=Never, 1=less than once per week, 2=once per week, 3=2-4 times/week, 4=nearly daily/daily, 5=greater than twice per day). Given intake for guideline 4 was assessed with only 1 item on the FFQ, the total guideline 4 score was the response to this single item (range 0-5), where higher scores indicate more frequently drinking sugar-sweetened drinks. This study used a factorial design, with 16 conditions (with ~4 participants) and was designed to collapse across conditions (i.e., comparing 8 conditions where factor is ON to 8 OFF conditions). Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 0, 10, 20 weeks
Population: as for outcome 17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | 2.07 (.31) | 2.21 (.30) | 2.07 (.31) | 2.16 (.29) | 2.04 (.30) | 2.19 (.30) | 2.24 (.29) | 2.00 (.31) | 2.12 (.21)
  20 weeks (post-treatment) | 1.29 (.28) | 1.11 (.27) | 1.29 (.28) | .96 (.26) | 1.28 (.28) | 1.28 (.28) | .94 (.27) | 1.31 (.28) | 1.12 (.19)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

32. Secondary Outcome: Treatment Acceptability: 10 Weeks
Description: An adapted 8- item version of the Treatment Acceptability Questionnaire (Hunsley, 1993) was used to assess intervention acceptability. Eight questions probed their program experience and how helpful/acceptable they found various intervention components (e.g., "How effective do you think this program is?"). Responses ranged from 1 = no/low acceptability to 7 = high acceptability. A total score was calculated as the average across all 8 items (range 8-56) where higher scores indicate greater treatment acceptability.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: 10 weeks (mid-treatment)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale | 47.51 (2.02) | 44.13 (1.97) | 46.25 (1.85) | 45.39 (2.03) | 44.87 (2.04) | 46.77 (1.89) | 44.82 (1.70) | 46.82 (2.09) | 45.76 (1.28)

33. Secondary Outcome: Treatment Acceptability: 20 Weeks
Description: as for outcome 32
Time Frame: 20 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale | 47.71 (2.11) | 46.46 (2.10) | 48.31 (1.94) | 45.87 (1.87) | 48.51 (2.21) | 45.67 (2.02) | 46.87 (1.53) | 47.31 (2.33) | 46.82 (1.25)

34. Secondary Outcome: Goals and Stages of Change- Household Member
Description: Two self-report items developed by the investigator assessed the goals of the selected household member at baseline: "On a scale of 1-100, how important is it that you adopt healthier eating habits right now?". Item 2 asked "On a scale of 1-100, how important is it that you help your household member adopt healthier eating habits right now?". For each item, household members responded on a scale from 0 - not important at all, 50 - about as important as most of the other things I would like to achieve now, to 100 - most important thing in my life now. Items were analyzed at individually, and each item ranged 0-100 where higher scores indicate higher importance of the associated goal.
Time Frame: 0 weeks
Population: Household members who served in a support role for participants assigned to the household support ON condition. We attempted to get data from all household members; however, only 17 responded on this item.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Household Condition: An adult household member attends one workshop session and three phone calls with the index participant. This household member receives weekly text messages for 20 weeks about program goals and ways to support the index participant.
  Household support: If participants are assigned to have household support ON, one adult in the household will receive weekly text messages designed to elicit support for changing food purchases. In addition, the index participant and household member will be invited to participate in one extra workshop session and three brief coaching calls focused on household support. If participants are assigned to have this OFF, household members will have no program involvement.
Arm/Group | Household Condition
Number analyzed (Participants) | 17
score on a scale
  Importance of Change Own Habits | 69.76 (19.94)
  Importance of Helping Participant Change Habits | 73.88 (22.32)

35. Secondary Outcome: Dietary Intake-household Member
Description: Household members completed the same 13-item Food Frequency Questionnaire as the index participant (adapted from Rifas-Shiman et al., 2001) to measure dietary intake. Household members are presented with 13 categories of foods that are relevant for each of the cancer prevention dietary guidelines (e.g., "Fresh, frozen, or canned fruit (not dried or fruit juice)", "Red meats such as beef, pork, lamb"). They rated how frequently they consume each category during an average week over the past month. Scale is as follows: 0 = Never, 1 = less than per week, 2= once per week, 3 = 2-4 times per week, 4 = nearly daily or daily, 5 = greater than twice per day. The 13 items are then classified into the guideline they pertain to and total guidelines scores were calculated as the average of responses to all relevant items (range 0-5) where higher scores indicate more frequently eating items associated with that nutrition guideline.
Time Frame: 0, 20 weeks
Population: Household members (among partners in the household condition). Household members who served in a support role for participants assigned to the household support ON condition. We attempted to get data from all household members; however, only 17 responded to this item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 17
score on a scale
  Guideline 1 (Baseline) | 2.78 (.83)
  Guideline 1 (Posttreatment) | 3.29 (.65)
  Guideline 2 (Baseline) | 2.49 (.72)
  Guideline 2 (Posttreatment) | 1.73 (.70)
  Guideline 3 (Baseline) | 2.24 (.66)
  Guideline 3 (Posttreatment) | 1.79 (.97)
  Guideline 4 (Baseline) | 1.65 (1.80)
  Guideline 4 (Posttreatment) | 1.41 (1.18)
Statistical Analysis 1: Comparison: Household Support - ON; Test type: Superiority; p < .05, t-test, 2 sided; Paired Sample T-test

36. Secondary Outcome: Treatment Acceptability - Household
Description: Household members completed the same adapted 8- item version of the Treatment Acceptability Questionnaire (Hunsley, 1993) as index participants. This measured acceptability of the intervention. Household members were presented with 8 questions about their experience during the program and how helpful/acceptable they found various intervention components to be (e.g., "How effective do you think this program is?", "How trustworthy do you think your coach was?". Household members responded to each question on a 7-point Likert scale where 1 = no/low acceptability and 7 = high acceptability. A total score was calculated as the average across all 8 items (range 8-56) where higher scores indicate greater treatment acceptability.
Time Frame: 20 weeks
Population: Household members (among partners in the household condition). Household members who served in a support role for participants assigned to the household support ON condition. We attempted to get data from all household members; however, only 17 responded on this item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 17
score on a scale | 45.00 (5.71)

37. Secondary Outcome: Dietary Intake- Household Member - FFQ (Guideline 1)
Description: Household members completed the same 13-item Food Frequency Questionnaire as the index participant (adapted from Rifas-Shiman et al., 2001) to measure dietary intake. To measure intake consistent with guideline 1 of the dietary cancer prevention guidelines (i.e., intake of fruits, vegetables, whole grains, and bean/ legumes ), household members rated how frequently they consumed these categories (4 items) during an average week over the past month. Scale was as follows: 0 = Never, 1 = less than once per week, 2= once per week, 3 = 2-4 times per week, 4 = nearly daily or daily, 5 = greater than twice per day. A total guideline 1 score was calculated as the average of responses to the 4 items (range 0-5), where higher scores indicate more frequently eating fruits, vegetables, whole grains, and beans/legumes.
Time Frame: 0, 20 weeks
Population: Household members (among partners in the household condition). Only half of participants were asked to include a household member, and 12 of these household members successfully provided data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 12
score on a scale
  0 weeks (baseline) | 2.73 (.67)
  20 weeks (post-treatment) | 3.38 (.67)
Statistical Analysis 1: Comparison: Household Support - ON; Test type: Superiority; p = .006, t-test, 2 sided; Paired samples t-test

38. Secondary Outcome: Dietary Intake - Household Member - FFQ (Guideline 2)
Description: Household members completed the same 13-item Food Frequency Questionnaire as the index participant (adapted from Rifas-Shiman et al., 2001) to measure dietary intake. To measure intake consistent with guideline 2 of the dietary cancer prevention guidelines (i.e., intake of processed foods high in fat, starches, or sugars), household members rated how frequently they consumed foods that fell into these categories (6 items) during an average week over the past month. Scale was as follows: 0 = Never, 1 = less than once per week, 2= once per week, 3 = 2-4 times per week, 4 = nearly daily or daily, 5 = greater than twice per day. A total guideline 2 score was calculated as the average of responses to the 6 items (range 0-5), where higher scores indicate more frequently eating processed foods high in far, starches, and sugars.
Time Frame: 0, 20 weeks
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 12
score on a scale
  0 weeks (baseline) | 2.65 (.63)
  20 weeks (post-treatment) | 1.71 (.76)
Statistical Analysis 1: Comparison: Household Support - ON; Test type: Superiority; p < .001, t-test, 2 sided; Paired samples t-test

39. Secondary Outcome: Dietary Intake-household Member - FFQ (Guideline 3)
Description: Household members completed the same 13-item Food Frequency Questionnaire as the index participant (adapted from Rifas-Shiman et al., 2001) to measure dietary intake. To measure intake consistent with guideline 3 of the dietary cancer prevention guidelines (i.e., intake of red and processed meats), household members rated how frequently they consumed red meats and processed meats (2 items) during an average week over the past month. Scale was as follows: 0 = Never, 1 = less than once per week, 2= once per week, 3 = 2-4 times per week, 4 = nearly daily or daily, 5 = greater than twice per day. A total guideline 3 score was calculated as the average of responses to the 2 items (range 0-5), where higher scores indicate more frequently eating red and processed meats.
Time Frame: 0, 20 weeks
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 12
score on a scale
  0 weeks (baseline) | 2.17 (.75)
  20 weeks (post-treatment) | 1.67 (1.09)
Statistical Analysis 1: Comparison: Household Support - ON; Test type: Superiority; p = .220, t-test, 2 sided; Paired samples t-test

40. Secondary Outcome: Dietary Intake-household Member - FFQ - Guideline 4
Description: Household members completed the same 13-item Food Frequency Questionnaire as the index participant (adapted from Rifas-Shiman et al., 2001) to measure dietary intake. To measure intake consistent with guideline 4 of the dietary cancer prevention guidelines (i.e., intake of sugar sweetened beverages), household members rated how frequently they consumed sugar sweetened beverages (1 item) during an average week over the past month. Scale was as follows: 0 = Never, 1 = less than once per week, 2= once per week, 3 = 2-4 times per week, 4 = nearly daily or daily, 5 = greater than twice per day. A total guideline 4 score was calculated as the response to this item (range 0-5), where higher scores indicate more frequently drinking sugar sweetened beverages.
Time Frame: 0, 20 weeks
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Household Support - ON
Number analyzed (Participants) | 12
score on a scale
  0 weeks (baseline) | 1.75 (1.91)
  20 weeks (post-treatment) | 1.50 (1.31)
Statistical Analysis 1: Comparison: Household Support - ON; Test type: Superiority; p = .623, t-test, 2 sided; Paired samples t-test

41. Other Pre Specified Outcome: Adherence to AICR Cancer Prevention Guidelines: Guideline 1
Description: To calculate adherence to the NCI dietary recommendations for guideline 1 (fruits, vegetables, and fiber), the WCRF/AICR scoring method from Turati et al., 2020 was used. This method has pre-defined cutoff values for the recommended levels of intake for each nutrient that is expected to have clinical significance. Based on their self-reported levels of dietary intake for whole grains, beans, fruits, and vegetable consumption, participants receive adherence scores for each dietary domain of 0 (failure to meet recommendation), 0.5 (partially meeting recommended levels), or 1 (fully meeting recommended level of intake). Guideline 1 (fruits, vegetables, and fiber) total adherence score (range 0-1) was calculated as the average of adherence scores for whole grains, beans, fruits, and vegetable consumption.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: Through a factorial design, participants were randomly assigned to receive coach monitoring (ON/OFF), benefits of change (ON/OFF), location triggered messaging (ON/OFF), and household support (ON/OFF).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | .38 (.05) | .48 (.05) | .45 (.06) | .40 (.05) | .47 (.06) | .38 (.05) | .44 (.05) | .41 (.05) | .43 (.04)
  20 weeks (post-treatment) | .50 (.06) | .39 (.06) | .44 (.06) | .45 (.06) | .44 (.06) | .45 (.06) | .44 (.06) | .45 (.06) | .45 (.04)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .577, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

42. Other Pre Specified Outcome: Adherence to AICR Cancer Prevention Guidelines: Guideline 2
Description: To calculate adherence to the NCI dietary recommendations for guideline 2 (intake of processed foods), the WCRF/AICR scoring method from Turati et al., 2020 was used. This method has pre-defined cutoff values for the recommended levels of intake for each nutrient that is expected to have clinical significance. Based on their self-reported levels of intake of added sugar, saturated fat, and sodium in processed foods, participants receive adherence scores for each dietary domain of 0 (failure to meet recommendation), 0.5 (partially meeting recommended levels), or 1 (fully meeting recommended level of intake). Guideline 2 total adherence score (range 0-1) was calculated as the average of adherence scores for consumption of added sugar, saturated fat, and sodium in processed foods.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | .47 (.05) | .58 (.05) | .57 (.05) | .48 (.05) | .54 (.05) | .51 (.05) | .48 (.05) | .58 (.05) | .53 (.04)
  20 weeks (post-treatment) | .71 (.06) | .77 (.06) | .80 (.06) | .69 (.05) | .75 (.06) | .73 (.05) | .79 (.05) | .70 (.05) | .74 (.04)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

43. Other Pre Specified Outcome: Adherence to AICR Cancer Prevention Guidelines: Guideline 3
Description: To calculate adherence to the NCI dietary recommendations for guideline 3 (intake of red and processed meats), the WCRF/AICR scoring method from Turati et al., 2020 was used. This method has pre-defined cutoff values for the recommended levels of intake for each nutrient that is expected to have clinical significance. Based on their self-reported levels of intake of red and processed meats, participants receive adherence scores for each dietary domain of 0 (failure to meet recommendation), 0.5 (partially meeting recommended levels), or 1 (fully meeting recommended level of intake). Guideline 3 total adherence score (range 0-1) was calculated as the average of adherence scores for red and processed meat intake.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | .56 (.06) | .55 (.06) | .61 (.06) | .50 (.06) | .64 (.06) | 48 (.06) | .55 (.06) | .57 (.06) | .56 (.04)
  20 weeks (post-treatment) | .72 (.06) | .69 (.06) | .70 (.06) | .72 (.05) | .73 (.06) | .68 (.05) | .79 (.05) | .63 (.05) | .71 (.04)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p < .001, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

44. Other Pre Specified Outcome: Adherence to AICR Cancer Prevention Guidelines: Guideline 4
Description: To calculate adherence to the NCI dietary recommendations for guideline 4 (intake of sugar sweetened beverages), the WCRF/AICR scoring method from Turati et al., 2020 was used. This method has pre-defined cutoff values for the recommended levels of intake for each nutrient that is expected to have clinical significance. Based on their self-reported levels of intake of sugar sweetened beverages, participants receive an adherence score of 0 (failure to meet recommendation), 0.5 (partially meeting recommended levels), or 1 (fully meeting recommended level of intake). Guideline 4 total adherence score (range 0-1) was calculated as adherence score for intake of sugar sweetened beverages.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 41
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 30 | 32 | 31 | 31 | 62
score on a scale
  0 weeks (baseline) | .26 (.07) | .26 (.07) | .21 (.07) | .31 (.06) | .26 (.07) | .26 (.06) | .30 (.07) | .23 (.07) | .26 (.05)
  20 weeks (post-treatment) | .40 (.07) | .43 (.07) | .38 (.07) | .45 (.07) | .38 (.07) | .45 (.07) | .43 (.07) | .40 (.07) | .41 (.05)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .008, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

45. Other Pre Specified Outcome: Grocery Store Purchases - Fruit
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Fruit purchases were calculated by tabulating the percent of fruit purchases divided by total purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: Through a factorial design, participants were randomly assigned to receive coach monitoring (ON/OFF), benefits of change (ON/OFF), location triggered messaging (ON/OFF), and household support (ON/OFF).
  Ns are lower for grocery store purchasing outcome vs. others because the aim was exploratory, as the project was pilot testing the grocery store purchase data collection system. Many participants had missing data.
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 7.57 (2.55) | 6.49 (2.61) | 7.07 (1.44) | 6.99 (2.31) | 4.29 (2.83) | 9.77 (2.38) | 3.54 (1.57) | 10.52 (2.13) | 7.03 (1.41)
  20 weeks (post-treatment) | 10.61 (5.66) | 7.55 (5.79) | 8.18 (3.19) | 9.97 (5.12) | 7.19 (6.28) | 10.96 (5.27) | 9.13 (3.49) | 9.02 (4.73) | 9.08 (3.14)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .601, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated Measures ANOVA

46. Other Pre Specified Outcome: Grocery Store Purchases - Vegetables
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Vegetable purchases were calculated by tabulating the percent of fruit purchases divided by total purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 7 | 5 | 3 | 9 | 8 | 4 | 4 | 8 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 6.14 (5.29) | 19.82 (5.41) | 13.14 (2.98) | 12.83 (4.79) | 14.65 (5.87) | 11.32 (4.93) | 14.23 (3.26) | 11.74 (4.42) | 12.98 (2.93)
  20 weeks (post-treatment) | 14.40 (7.70) | 30.61 (7.87) | 22.60 (4.34) | 22.41 (6.97) | 28.57 (8.54) | 16.44 (7.17) | 22.61 (4.74) | 22.40 (6.43) | 22.51 (4.27)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .088, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

47. Other Pre Specified Outcome: Grocery Store Purchases - Meat
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Meat purchases were calculated by tabulating the percent of meat purchases divided by total purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 7 | 5 | 3 | 9 | 8 | 4 | 4 | 8 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 3.87 (2.83) | 7.48 (2.83) | 5.03 (1.60) | 6.32 (2.56) | 6.50 (3.14) | 4.86 (2.63) | 6.21 (1.74) | 5.14 (2.36) | 5.68 (1.57)
  20 weeks (post-treatment) | 9.25 (4.62) | 7.72 (4.73) | 7.32 (2.61) | 9.65 (4.18) | 6.83 (5.13) | 6.83 (5.13) | 10.07 (2.84) | 6.90 (3.86) | 8.48 (2.56)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .210, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

48. Other Pre Specified Outcome: Grocery Store Purchases - Grains and Beans
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Grains/beans purchases were calculated by tabulating the percent of grains and beans purchases divided by total purchases. Scores range from 0-100%.This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 11.28 (6.39) | 15.71 (6.54) | 8.75 (3.61) | 18.24 (5.78) | 16.47 (7.09) | 10.53 (5.95) | 15.78 (3.93) | 11.21 (5.34) | 13.50 (3.54)
  20 weeks (post-treatment) | 5.64 (2.65) | 5.53 (2.71) | 4.57 (1.50) | 6.60 (2.40) | 6.87 (2.94) | 4.30 (2.47) | 4.69 (1.63) | 6.48 (2.22) | 5.59 (1.47)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .060, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

49. Other Pre Specified Outcome: Grocery Store Purchases - Sugar-Sweetened Beverages
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Sugar-sweetened beverage (SSB) purchases were calculated by tabulating the percent of SSB purchases divided by total purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 9.88 (1.95) | 5.88 (1.99) | 6.92 (1.10) | 8.84 (1.76) | 7.64 (2.16) | 8.12 (1.81) | 7.43 (1.20) | 8.33 (1.63) | 7.88 (1.08)
  20 weeks (post-treatment) | 15.11 (5.25) | 5.52 (5.37) | 13.07 (2.96) | 7.56 (4.75) | 7.30 (5.83) | 13.32 (4.89) | 8.20 (3.23) | 12.43 (4.39) | 10.31 (2.91)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .370, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

50. Other Pre Specified Outcome: Grocery Store Purchases - Sweets
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Sweets purchases were calculated by tabulating the percent of meat purchases divided by total sweets purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 20.11 (5.83) | .00 (5.96) | 13.68 (3.29) | 6.43 (5.27) | 3.24 (6.47) | 16.87 (5.43) | 13.33 (3.59) | 6.78 (4.87) | 10.06 (3.23)
  20 weeks (post-treatment) | 10.71 (6.20) | 13.78 (6.33) | 13.89 (3.50) | 10.61 (5.60) | 19.80 (6.87) | 4.70 (5.77) | 14.22 (3.81) | 10.27 (5.17) | 12.25 (3.43)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .556, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated Measures ANOVA

51. Other Pre Specified Outcome: Grocery Store Purchases - Snacks
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Snack purchases were calculated by tabulating the percent of snack purchases divided by total purchases. Scores range from 0-100%.
  This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 13.37 (3.70) | 7.16 (3.79) | 10.56 (2.09) | 9.97 (3.35) | 11.70 (4.11) | 8.83 (3.45) | 9.72 (2.28) | 10.82 (3.09) | 10.27 (2.05)
  20 weeks (post-treatment) | 14.81 (4.22) | 5.11 (4.32) | 7.33 (2.38) | 12.59 (3.82) | 6.30 (4.69) | 13.61 (3.93) | 8.22 (2.60) | 11.69 (3.53) | 9.96 (2.34)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .913, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated measures ANOVA

52. Other Pre Specified Outcome: Grocery Store Purchases - Other Processed Foods
Description: To measure grocery purchasing, an API transferred participants' item-level food purchases to the study database whenever they shopped at designated grocery stores (Wegmans, ShopRite, Target, and Walmart). Each item in the shopping trip was linked to an existing nutrition databases (e.g., FNDDS) to categorize it into a NCI relevant category and to pull nutritional information. Processed food purchases were calculated by tabulating the percent of processed food purchases divided by total purchases. Scores range from 0-100%.This pilot study used a factorial design, with 16 conditions and typically 4 participants per condition. The study was designed with the intent to collapse across conditions for all analyses, such that the 8 conditions in which a given factor is ON would be compared to the 8 conditions in which that factor was OFF. Participants are counted multiple times in the table, such that the total number of participants in any ON/OFF condition pair will equal the full sample.
Time Frame: Baseline and post-treatment (0 and 20 weeks)
Population: as for outcome 45
Measure: Mean (Standard Error); unit: percentage of grocery store purchases
Arm/Group | Coach Monitoring - ON | Coach Monitoring - OFF | Benefits of Change - ON | Benefits of Change - OFF | Location Triggered Messaging - ON | Location-Triggered Messaging - OFF | Household Support - ON | Household Support - OFF | Full Sample
Number analyzed (Participants) | 5 | 7 | 9 | 3 | 4 | 8 | 8 | 4 | 12
percentage of grocery store purchases
  0 weeks (baseline) | 27.78 (9.50) | 37.45 (9.72) | 34.84 (5.36) | 30.40 (8.60) | 35.52 (10.55) | 29.71 (8.85) | 29.76 (5.85) | 35.47 (7.94) | 32.62 (5.26)
  20 weeks (post-treatment) | 19.48 (9.86) | 24.19 (10.08) | 23.06 (5.56) | 20.62 (8.92) | 17.14 (10.94) | 26.53 (9.18) | 22.86 (6.07) | 20.81 (8.32) | 21.84 (5.46)
Statistical Analysis 1: Comparison: Full Sample; Test type: Superiority; p = .241, ANOVA — The reported p-value reflects the change across time for the full sample; Repeated Measures ANOVA

ADVERSE EVENTS:
Time Frame: Pre-treatment to post-treatment (20 weeks)
Groups:
- Condition 14: Location triggered messaging - OFF, Benefits of change - OFF, Coach monitoring - ON, Household support - OFF.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/2 | 0/2 | 0/7 | 0/2 | 0/5 | 0/2 | 0/3 | 0/5 | 0/6 | 0/2 | 0/5 | 0/2 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/2 | 0/2 | 0/7 | 0/2 | 1/5 | 0/2 | 0/3 | 0/5 | 0/6 | 0/2 | 0/5 | 0/2 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/2 | 0/2 | 0/7 | 0/2 | 0/5 | 0/2 | 0/3 | 0/5 | 0/6 | 0/2 | 0/5 | 0/2 | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=4) | Condition 2 (N=7) | Condition 3 (N=2) | Condition 4 (N=2) | Condition 5 (N=7) | Condition 6 (N=2) | Condition 7 (N=5) | Condition 8 (N=2) | Condition 9 (N=3) | Condition 10 (N=5) | Condition 11 (N=6) | Condition 12 (N=2) | Condition 13 (N=5) | Condition 14 (N=2) | Condition 15 (N=4) | Condition 16 (N=4)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant was hospitalized for 4 weeks due to an infection unrelated to the study. The participant recovered from the infection with antibiotics.

LIMITATIONS AND CAVEATS:
Challenges with reliability of geofencing (location-triggered messages) and passive collection of purchasing data. Purchases monitored from only select stores and not other outlets (e.g., farmer's markets). Purchasing behavior does not fully align with consumption (e.g., individuals purchase items at the store for others). Sample characteristics limit generalizability. Different dietary intake assessments (ASA24 was high burden). No control condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04947150/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04947150/SAP_002.pdf
  • Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04947150/ICF_000.pdf